CLINICAL TRIAL: NCT00127946
Title: Randomized Trial of AMNIOECHANGE in Gastroschisis Affected Foetuses
Brief Title: Trial of AMNIOECHANGE in Gastroschisis Affected Foetuses
Acronym: AMNIOECHANGE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Saliha DJANE, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P040416
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2005-08

CONDITIONS: Gastroschisis
MeSH Terms: conditions — Gastroschisis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMNIOECHANGE (Active Comparator): The AMNIOECHANGE consists of a transabdominal infusion of saline.They will be repeated every 15 days from 30 week of amenorrhea.
  Interventions: Procedure: AMNIOECHANGE
- placebo (No Intervention): This will be done at the same place and under the same aseptic conditions a AMNIOECHANGE true.
  Interventions: Procedure: AMNIOECHANGE

INTERVENTIONS:
Procedure: AMNIOECHANGE — The AMNIOECHANGE consists of a transabdominal infusion of saline (heated to 37 ° C) with a needle 18 or 20 gauge under ultrasound monitoring while avoiding the placenta. In the case of a normal amniotic fluid, it must be replaced volume per volume of saline (eg depending on the tank where the puncture is made, it can be 300 per 300 ml). The total amount of amniotic fluid exchange is 600-900 ml. In cases of oligohydramnios, the AMNIOECHANGE results in a normalized volume of amniotic fluid.

SUMMARY:
Hypothesis: Gastroschisis is a localised disruption of the abdominal layer. It occurs early in gestation, and the bowel is therefore bathing in the amniotic fluid and can be constricted at the level of the abdominal hole. The bowel is therefore submitted to different injuries partly attributable to the contact with amniotic fluid contaminated by digestive compounds and inducing an inflammatory reaction. Experimental studies on animal models and preliminary data in humans indicate that changing regularly the amniotic fluid (i.e. AMNIOECHANGE) would improve the outcome of theses fetuses and then neonates.

DETAILED DESCRIPTION:
Primary Objective: To compare prospectively the effect of AMNIOECHANGE against classical care on the delay of full enteral feeding in gastroschisis affected foetuses

Study:

* Multicenter, Randomized.
* Inclusion at 20 GA (gestational age) weeks.
* AMNIOECHANGE every 2 weeks from 30 GA weeks

Subject: 140 inclusion during 3 years

Analysis: Triangular Sequential Evaluation

ELIGIBILITY:
Inclusion Criteria:

* Seen before 30 GA weeks
* Normal karyotype
* Single pregnancy
* Isolated gastroschisis
* No associated disease (maternal)
* Accept randomization and understand the study

Exclusion Criteria:

* Maternal diabetes
* Maternal infection with HIV, hepatitis
* Preexistent oligohydramnios before inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2005-11; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Duration of ventilation in the ICU and the duration of parenteral nutrition | 7 days and 45 days after the birth of the child
  The primary outcome was a composite endpoint based on the duration of ventilation in the ICU and the duration of parenteral nutrition

SECONDARY OUTCOMES:
Evaluation of the contribution of iterative AMNIOECHANGE | 7 days, 45 days, 12 months and 18 months
  * Obstetric complications: chorioamnionitis, preterm labor, premature rupture of membranes,
  * Aspect périviscérite, age out of intensive care and the initialization of enteral nutrition, infection
  * Evaluation of complications of surgery, duration of hospitalization.
  * And to determine prenatal prognostic factors: 1. Ultrasound 2. Biological and postnatal: Histology

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Luton, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre hospital, AP-HP, Paris, Paris, France

REFERENCES:
- [Derived] Luton D, Mitanchez D, Winer N, Muller F, Gallot D, Perrotin F, Jouannic JM, Bretelle F, de Lagausie P, Ville Y, Guibourdenche J, Oury JF, Alberti C, Benachi A. A randomised controlled trial of amnioexchange for fetal gastroschisis. BJOG. 2019 Sep;126(10):1233-1241. doi: 10.1111/1471-0528.15804. Epub 2019 May 20. PMID 31033140